CLINICAL TRIAL: NCT04513379
Title: Efficacy and Safety of 400 mg Efavirenz Versus Standard 600 mg Dose in HIV/TB Co-infected Patients Receiving Rifampicin Based Anti-TB Therapy
Brief Title: Efficacy of 400 mg Efavirenz Versus Standard 600 mg Dose in HIV/TB Co-infected Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Public Health Clinical Center (Other Government)
Responsible Party: Principal Investigator, Jun Chen, Shanghai Public Health Clinical Center, Shanghai Public Health Clinical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EDOSE
Record Dates: First submitted 2020-08-12; First posted 2020-08-14 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: HIV Infections; Tuberculosis
MeSH Terms: conditions — HIV Infections; Tuberculosis | interventions — efavirenz

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Trial (Experimental): EFV 400mg
  Interventions: Drug: Efavirenz 400mg
- Control (Active Comparator): EFV 600mg
  Interventions: Drug: Efavirenz 600mg

INTERVENTIONS:
Drug: Efavirenz 600mg — EFV 600 mg per day given orally
  Arms: Control
Drug: Efavirenz 400mg — 2 tablets of EFV 200 mg per day given orally
  Arms: Trial

SUMMARY:
TB is the most common cause of death in patients with HIV worldwide. Rifampicin [RIF] is the cornerstone of anti-TB therapy. Current guideline recommend efavirenz (EFV) 600mg per day as the first of choice for HIV/TB co-infection. Co-administration of EFV with RIF decrease the plasma concentration of EFV. Because of better safety profiles, EFV 400mg has replaced the EFV 600mg as the first-line antiretroviral therapy in people living with HIV. However, the efficacy of EFV 400mg when co-administrated with RIF in HIV/TB co-infection is unclear. This study is designed to evaluate the efficacy and safety of EFV 400mg versus EFV 600mg in HIV/TB co-infected patients receiving RIF based anti-TB therapy.

ELIGIBILITY:
Inclusion Criteria:

* Subject or the subject's legal representative is willing and able to understand and provide signed and dated written informed consent prior to Screening
* Adult subject (at least 18 years of age)
* Naive to antiretroviral therapy (<=14 days of prior therapy with any antiretroviral drug following a diagnosis of HIV-1 infection)
* CD4+ cell count is >= 50 cells/ cubic millimetre (mm^3) at Screening
* A female subject may be eligible to enter and participate in the study if she: is of non-childbearing potential defined as either postmenopausal (12 months of spontaneous amenorrhea and >=45 years of age) or physically incapable of becoming pregnant or does not want to pregnancy
* New diagnosis of TB (microbiology or molecular methods or clinical diagnosis) and started rifampicin based regimen for less no longer than 8 weeks at screening

Exclusion Criteria:

* Evidence of RIF resistance of Mycobacterium tuberculosis either by culture or validated nucleic acid amplification test
* Concomitant disorders or conditions for which isoniazid, RIF, pyrazinamide, or ethambutol are contraindicated
* Central nervous system TB
* Women who are pregnant or breastfeeding
* Subjects with moderate to severe hepatic impairment (Class B or C) as determined by Child-Pugh classification unstable liver disease
* Anticipated need for hepatitis C virus (HCV) therapy during the study period
* History or presence of allergy or intolerance to the study drugs or their components or drugs of their class
* Subjects who, in the investigator's judgment, pose a significant suicidality risk.
* Treatment with any of the following agents within 28 days of Screening: radiation therapy, cytotoxic chemotherapeutic agents, any immunomodulators that alter immune response
* Exposure to an experimental drug or experimental vaccine within either 28 days, 5 half-lives of the test agent, or twice the duration of the biological effect of the test agent, whichever is longer, prior to the first dose of investigate drug
* Any evidence of primary viral resistance to Nucleoside reverse transcriptase inhibitor (NRTIs), Non-nucleoside reverse transcriptase inhibitor (NNRTIs) based on the presence of any major resistance-associated mutation in the Screening result or, if known, any historical resistance test result.
* Any acute laboratory abnormality at Screening, which, in the opinion of the investigator, would preclude the subject's participation in the study of an investigational compound.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2022-10-30 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Plasma HIV-1 RNA < 50 Copies/Milliliter at Week 48 Using the US Food and Drug Administration (FDA) Snapshot Algorithm | Week 48
  The percentage of participants who were responders was assessed at the study Week 48 for participants randomized to receive at least one dose of study medication. Response was assessed using a modified FDA Snapshot algorithm

SECONDARY OUTCOMES:
Percentage of Participants With Plasma HIV-1 RNA < 50 Copies/Milliliter at Week24 Using the US Food and Drug Administration (FDA) Snapshot Algorithm | Week 24
  The percentage of participants who were responders was assessed at the study Week 24 for participants randomized to receive at least one dose of study medication. Response was assessed using a modified FDA Snapshot algorithm
Percentage of Participants Without Confirmed Virologic Withdrawal and Without Discontinuation Due to Treatment-related Reasons at Week 24 and Week 48 | Week 24 and Week 48
  Percentage of participants not meeting confirmed virologic withdrawal criteria nor discontinued due to treatment related reasons at the time of analysis at Week 24 (through Day 210) and Week 48 (through Day 350) is presented by treatment group.
Number of Participants With Tuberculosis (TB) Associated Immune Reconstitution Inflammatory Syndrome (IRIS) | Week 12
  Participants were monitored for signs and symptoms of TB-IRIS. Participants with IRIS symptoms in any adverse events or HIV associated. conditions were classified by the study investigators in the following categories as met criteria for TB-IRIS, possibly met criteria for TB-IRIS and suspected TB-IRIS but not possible to adjudicate.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Chen, M.D, Principal Investigator — Shanghai Public Health Clinical Center